CLINICAL TRIAL: NCT05615220
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized Withdrawal Study to Evaluate the Safety and Maintenance of Efficacy of Ecopipam in Children, Adolescents and Adults With Tourette's Disorder
Brief Title: Ecopipam Tablets to Study Tourette's Disorder in Children, Adolescents and Adults
Acronym: D1AMOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EBS-101-TD-301; 2023-503494-38-00 (EU CTIS Number); 2022-001961-11 (EudraCT Number)
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-04

CONDITIONS: Tourette Disorder
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Intervention Model Description: Sequential Assignment This is a multicenter study which includes an open-label period followed by double-blind, placebo-controlled, randomized withdrawal period.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This includes an open-label period followed by a double-blind, placebo-controlled, randomized withdrawal period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1.8 mg/kg/day ecopipam (2 mg/kg/day ecopipam HCl) (Experimental): Ecopipam 11.2, 22.4, 33.6, 44.8, 67.2 and 89.6 mg tablets (containing 12.5, 25, 37.5, 50, 75 and 100 mg ecopipam HCl, respectively); 1.8 mg/kg/day ecopipam (2 mg/kg/day ecopipam HCl) target dose; oral administration daily in evenings.
  Interventions: Drug: Ecopipam Hydrochloride
- Placebo during R/WD Phase (Placebo Comparator): Matching Placebo tablets during R/WD period taken orally in the evening.
  Interventions: Drug: Ecopipam Hydrochloride

INTERVENTIONS:
Drug: Ecopipam Hydrochloride — Selective dopamine D1 and D5 receptor antagonist

SUMMARY:
This Phase 3 multicenter study evaluates the maintenance of efficacy, safety and tolerability of ecopipam tablets in children, adolescents and adults in the treatment of Tourette's Disorder (TD). The study includes an open-label period followed by a double-blind, placebo-controlled, randomized withdrawal period.

DETAILED DESCRIPTION:
Following a 28-day Screening period and Baseline visit, eligible subjects will be enrolled into the open-label Stabilization period comprised of a 4-week Titration phase to achieve a target steady-state dose of 1.8 mg/kg/day ecopipam (2 mg/kg/day ecopipam HCl) followed by an 8-week open-label Maintenance phase. Responders to ecopipam will be randomized to ecopipam 1.8 mg/kg/day (2 mg/kg/day ecopipam HCl) or placebo in a 1:1 fashion and enter the double-blind Randomized-Withdrawal (R/WD) period at Week 12. During the 12-week R/WD period, any subject meeting Relapse criteria will be withdrawn from blinded study medication and complete end of study assessments including safety follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 years of age
* ≥ 18 kg (~ 40 lbs.)
* TD diagnosis and both motor and vocal tics that cause impairment with normal routines
* Minimum score of 20 on the YGTSS-R Total Tic Score
* May not be taking any medications used to treat motor or vocal tics for at least 14 days prior to Baseline.
* Effective contraception during the study and 30 days after last study dose for sexually active subjects

Exclusion Criteria:

* Previous exposure to ecopipam
* Certain mood or psychiatric disorders (i.e., dementia, bipolar disorder, schizophrenia, major depressive disorder)
* Unstable medical illness or clinically significant lab abnormalities
* Risk of suicide
* Pregnant or lactating women
* Moderate to severe renal insufficiency
* Hepatic insufficiency
* Positive urine drug screen
* Unstable doses for drugs to treat anxiety, depression, Attention Deficit Hyperactivity Disorder
* Certain medications that would lead to drug interactions
* Recent behavioral therapy

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (56):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - CenExel CIT-IE, Bellflower, California
  - Cortica Site Network, Glendale, California
  - Amnova Clinical Research, Irvine, California
  - Cortica Site Network - San Rafael, San Rafael, California
  - Syrentis Clinical Research, Santa Ana, California
  - Yale School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Research in Miami Inc, Hialeah, Florida
  - Emcrown Clinical Research, Jensen Beach, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Florida International Research Center, Miami, Florida
  - Care Research Center, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - APG Research LLC, Orlando, Florida
  - University of South Florida, St. Petersburg, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Jedidiah Clinical Research, Tampa, Florida
  - Pediatric Neurology, PA, Winter Park, Florida
  - Advanced Discovery Research, LLC, Atlanta, Georgia
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Atlanta Behavioral Research, LLC., Atlanta, Georgia
  - Lurie Children Hospital of Chicago, Chicago, Illinois
  - 1725 W. Harrison St., Suite 755, Chicago, Illinois
  - The University of Chicago Hospitals, Chicago, Illinois
  - Josephson-Wallack-Munshower Neurology, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Umass Chan Medical School, Worcester, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Midwest Research Group, Saint Charles, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Alivation Research, Lincoln, Nebraska
  - NYU Child Study Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wake Forest Baptist Medical Center - PPDS, Winston-Salem, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Coastal Pediatric Research, Charleston, South Carolina
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital (TCH), Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Perceptive Pharma Research (PPR), Richmond, Texas
  - Road Runner Research Ltd., San Antonio, Texas
  - Cedar Clinical Research, Draper, Utah
  - Core Clinical Research, Everett, Washington
- Bulgaria (4):
  - Center Spectar-Plovdiv, Plovdiv, Bulgaria
  - ASMP-IP- d-r Kayryakova, Sofia, Sofia-Grad
  - Kalimat Medical Center_Sofia, Sofia
  - DCC Mladost-M Varna, Varna
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - The Kids Clinic Inc, Ajax, Ontario
- Borne og Ungeafdelingen, Herlev, Denmark
- France (3):
  - CHU Grenoble Alpes - Hopital Couple Enfant, Grenoble
  - Hôpital Fondation Rothschild, Paris
  - CHU Strasbourg-Hopital de Hautepierre, Strasbourg
- Germany (3):
  - Psychiatric Clinic of Ludwig Maximilians Universitaet Muenchen, Munich, Bavaria
  - Department of Psychiatry, Socialpsychiatry and Psychotherapy, Hannover Medical School, Hanover, Lower Saxony
  - Zentralinstitut fuer Seelische Gesundheit, Mannheim, Mannheim
- Hungary (3):
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar Gyermek, Szeged, Csongrád megye
  - Vadaskert Gyermek- es Ifjusagpszichiatriai Korhaz es Szakambulancia, Budapest
  - Bethesda Childrens Hospital(Magyarországi Református Egyház Bethesda Gyermekkórháza), Budapest
- Italy (6):
  - Istituto Di Ricovero E Cura A Carattere Scientifico IRCCS Eugenio Medea, Bosisio Parini, LC
  - IRCCS Istituto Neurologico Carlo Besta, Milan, Milano
  - Universita degli Studi di Napoli Federico II, Napoli, Napoli
  - Ospedale Pediatrico Bambino Gesù, Roma, RM
  - Azienda Ospedaliera Vittorio Emanuele Policlinico // Azienda Ospedaliera Policlinico San Marco, Catania
  - Ospedale Pediatrico Istituto Giannina Gaslini di Genova, Genova
- Poland (5):
  - Clinical Research Center Sp. z o.o. MEDIC-R Sp.k., Poznan, Poland
  - Gdanskie Centrum Zdrowia Sp z o.o., Gdansk, Pomeranian Voivodeship
  - Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice, Silesian Voivodeship
  - Wojewdzki Specjalistyczny Szpital Dziecicy im. sw. Ludwika w Krakowie, Krakow, Woj. Malopolskie
  - Centrum Medyczne Plejady, Krakow
- Spitalul Clinic de Psihiatrie Prof Dr Al. Obregia Bucureti, Dorobanți, Romania
- Serbia (4):
  - Institute of Mental Health, Belgrade, Belgrad
  - Clinical Centre Nis Center of Mental Health, Niš, Serbia
  - Clinical Center Vojvodina, Novi Sad, Serbia
  - Clinic of Neurology and Psychiatry for Children and Adolescents, Belgrade
- Spain (7):
  - Hospital Universitario Fundacion Alcorcon HUFA, Alcorcón, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen del Rocío, C/Antonio Maura Montaner, s/n, edificio IBiS, Seville, Sevilla
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Virgen Macarena Unidad de Investigacion Neurologia, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The multicenter study was conducted globally in the United States, Bulgaria, Canada, Denmark, France, Germany, Hungary, Italy, Poland, Romania, Serbia, and Spain from 31 January 2023 to 04-February 2025.
Pre-assignment Details: Participants with a diagnosis of Tourette's Disorder were enrolled in this study to receive oral ecopipam in an Open-label Stabilization Period and a Double-blind Randomized Withdrawal (R/WD) Period and then followed for safety up to 30 days post-last dose.
Groups:
- Open-label stabilization Period: Ecopipam 1.8 mg/kg/day: All participants in the open-label stabilization period received a target steady-state dose of 1.8 milligram per kilogram per day (mg/kg/day) ecopipam (2 mg/kg/day ecopipam hydrochloride [HCl]) tablets based on body weight, administered orally, once daily in the evening during a 4-week titration phase and further followed by an 8-week maintenance phase.
- Double-blind R/WD Period: Ecopipam 1.8 mg/kg/day: Participants who met stabilization criteria were randomized to receive ecopipam 1.8 mg/kg/day (ecopipam HCl 2 mg/kg/day) orally once daily in the evening, up to 12 weeks in Double-blind R/WD Phase.
- Double-blind R/WD Period: Placebo: Participants received matching placebo tablets, once daily, up to 12 weeks in Double-blind R/WD Phase. Participants randomized to placebo were tapered off ecopipam in a blinded fashion, in decrements of 22.4 milligrams per day (mg/day) (25 mg/day ecopipam HCl).
Period: Open label stabilization Part (12 weeks)
Arm/Group | Open-label stabilization Period: Ecopipam 1.8 mg/kg/day | Double-blind R/WD Period: Ecopipam 1.8 mg/kg/day | Double-blind R/WD Period: Placebo
Started | 216 | 0 | 0
Completed | 104 | 0 | 0
Not Completed | 112 | 0 | 0
Not completed — Failure to meet responder criteria | 36 | 0 | 0
Not completed — Study end once relapsed goal met | 21 | 0 | 0
Not completed — Adverse Event | 33 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Other | 6 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0
Period: Double Blind R/WD Part (12-24 weeks)
Arm/Group | Open-label stabilization Period: Ecopipam 1.8 mg/kg/day | Double-blind R/WD Period: Ecopipam 1.8 mg/kg/day | Double-blind R/WD Period: Placebo
Started | 0 | 51 (All participants (Responders) to ecopipam in the open-label Stabilization period were randomized 1:1 to either ecopipam or matching placebo for the R/WD period.) | 53 (All participants (Responders) to ecopipam in the open-label Stabilization period were randomized 1:1 to either ecopipam or matching placebo for the R/WD period.)
Completed | 0 | 21 | 13
Not Completed | 0 | 30 | 40
Not completed — Relapsed | 0 | 21 | 36
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Study end once relapsed goal met | 0 | 6 | 2
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Open-label Stabilization Period: Ecopipam 1.8 mg/kg/Day: All participants in the open-label stabilization period who received a target steady-state dose of 1.8 mg/kg/day ecopipam (2 mg/kg/day ecopipam hydrochloride [HCl]) tablets based on body weight, administered orally, once daily in the evening during a 4-week titration phase and further followed by an 8-week maintenance phase.
Arm/Group | Open-label Stabilization Period: Ecopipam 1.8 mg/kg/Day
Number analyzed (Participants) | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 186
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 7
  White | 196
  More than one race | 4
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Relapse in Participants Greater Than and Equal to (>=) 6 and Less Than (<) 18 Years During the Double-Blind R/WD
Description: Time to relapse defined as a loss of >=50 percent (%) of the improvement experienced on the Yale Global Tic Severity Scale-Total Tic Score (YGTSS-TTS) from Baseline to the last visit in the Open-Label Stabilization Period (Week 12), or initiation of additional medications to treat symptoms of Tourette's Disorder (TD), or requirement of hospitalization for worsening symptoms of TD in participants between the ages of >= 6 and <18 years for ecopipam compared to those receiving placebo during the double-blind, R/WD period. The YGTSS was a clinician-completed rating scale used to quantify overall tic severity in participants with TD as well as specific subdomains of tic number, frequency, intensity, complexity and interference. Each of these subdomains was scored, on a 0 to 5 scale, separately for motor and vocal tics and then summed across both motor and vocal tics to yield a total tic score ranging from 0 to 50. Higher scores represented more severe symptoms.
Time Frame: From randomization at Week 12 through the end of the double-blind R/WD period (up to Week 24)
Population: The modified intention-to-treat (mITT) set included all randomized participants who received at least 1 dose of study drug post-randomization.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Double- Blind R/WD Period: Ecopipam 1.8 mg/kg/Day: Participants who met stabilization criteria were randomized to receive ecopipam 1.8 mg/kg/day (ecopipam HCl 2 mg/kg/day) orally once daily in the evening, up to 12 weeks in Double-Blind R/WD Phase.
- Double- Blind R/WD Period: Placebo: Participants received matching placebo tablets, once daily, up to 12 weeks in Double-blind R/WD Phase. Participants randomized to placebo were tapered off ecopipam in a blinded fashion, in decrements of 22.4 milligrams per day (mg/day) (25 mg/day ecopipam HCl).
Arm/Group | Double- Blind R/WD Period: Ecopipam 1.8 mg/kg/Day | Double- Blind R/WD Period: Placebo
Number analyzed (Participants) | 43 | 47
weeks | NA [4.1 to NA] — Here "NA" means median and upper limit of 95% confidence interval could not be estimated due to insufficient events within the treatment group. | 4.0 [2.4 to 6.1]

2. Secondary Outcome: Time From Randomization to Relapse in All Participants During the Double-Blind R/WD Period
Description: Time From Randomization (Week 12) to relapse defined as a loss of >= 50% of the improvement experienced on the YGTSS-TTS from Baseline to the last visit in the Open-Label Stabilization Period (Week 12), or initiation of additional medications to treat symptoms of TD, or requirement of hospitalization for worsening symptoms of TD in all participants during the Double-Blind R/WD period for ecopipam compared to placebo. The YGTSS was a clinician-completed rating scale used to quantify overall tic severity in children and adults with TD as well as specific subdomains of tic number, frequency, intensity, complexity and interference. Each of these subdomains was scored, on a 0 to 5 scale, separately for motor and vocal tics and then summed across both motor and vocal tics to yield a total tic score ranging from 0 to 50. Higher scores represented more severe symptoms.
Time Frame: From randomization at Week 12 through the end of the double-blind R/WD period (up to Week 24)
Population: The mITT Set included all randomized participants who received at least 1 dose of study drug post-randomization.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Double- Blind R/WD Period: Ecopipam 1.8 mg/kg/Day: Participants who met stabilization criteria were randomized to receive ecopipam 1.8 mg/kg/day (ecopipam HCl 2 mg/kg/day) orally OD in the evening, up to 12 weeks in Double-Blind R/WD Phase.
Arm/Group | Double- Blind R/WD Period: Ecopipam 1.8 mg/kg/Day | Double- Blind R/WD Period: Placebo
Number analyzed (Participants) | 51 | 53
weeks | NA [4.1 to NA] — Here "NA" means median and upper limit of 95% confidence interval could not be estimated due to insufficient events within the treatment group. | 4.0 [2.4 to 6.1]

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to end of double blind follow up period (up to Day 199)
Description: Safety Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Open-label Stabilization Period: Ecopipam 1.8 mg/kg/Day: All participants in the open-label stabilization period were received a target steady-state dose of 1.8 mg/kg/day ecopipam (2 mg/kg/day ecopipam hydrochloride [HCl]) tablets based on body weight, administered orally, once daily in the evening during a 4-week titration phase and further followed by an 8-week maintenance phase.
- Double- Blind R/WD Period: Placebo: Participants received matching placebo tablets, once daily, up to 12 weeks in Double-blind R/WD Phase. Participants randomized to placebo were tapered off ecopipam in a blinded fashion, in decrements of 22.4 mg/day (25 mg/day ecopipam HCl).
Arm/Group | Open-label Stabilization Period: Ecopipam 1.8 mg/kg/Day | Double-blind R/WD Period: Ecopipam 1.8 mg/kg/Day | Double- Blind R/WD Period: Placebo
All-Cause Mortality (participants affected / at risk) | 0/216 | 0/51 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/216 | 1/51 | 2/53
Other Adverse Events (participants affected / at risk) | 140/216 | 20/51 | 22/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Stabilization Period: Ecopipam 1.8 mg/kg/Day (N=216) | Double-blind R/WD Period: Ecopipam 1.8 mg/kg/Day (N=51) | Double- Blind R/WD Period: Placebo (N=53)
Tourette's disorder (Congenital, familial and genetic disorders) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Stabilization Period: Ecopipam 1.8 mg/kg/Day (N=216) | Double-blind R/WD Period: Ecopipam 1.8 mg/kg/Day (N=51) | Double- Blind R/WD Period: Placebo (N=53)
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 14 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 1
Influenza like illness (General disorders) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 3 | 0
Nasopharyngitis (Infections and infestations) | 5 | 0 | 2
Bronchitis (Infections and infestations) | 4 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 3 | 1 | 0
Influenza (Infections and infestations) | 2 | 1 | 0
Viral infection (Infections and infestations) | 2 | 1 | 0
Ear infection (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 1
Acute sinusitis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 0
Blood glucose increased (Investigations) | 1 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 24 | 0 | 0
Headache (Nervous system disorders) | 19 | 2 | 3
Dizziness (Nervous system disorders) | 2 | 1 | 0
Migraine (Nervous system disorders) | 1 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 20 | 1 | 1
Insomnia (Psychiatric disorders) | 16 | 3 | 5
Tic (Psychiatric disorders) | 15 | 2 | 1
Depressed mood (Psychiatric disorders) | 8 | 0 | 1
Irritability (Psychiatric disorders) | 6 | 1 | 0
Restlessness (Psychiatric disorders) | 5 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 5 | 0 | 1
Agitation (Psychiatric disorders) | 2 | 2 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1 | 3
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT05615220/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT05615220/SAP_001.pdf